CLINICAL TRIAL: NCT02914457
Title: Left Ventricular Synchronous Versus Sequential MultiSpot Pacing for CRT
Brief Title: Left Ventricular Synchronous Versus Sequential MultiSpot Pacing for Cardiac Resynchronization Therapy (CRT)
Acronym: SYNSEQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYNSEQ
Record Dates: First submitted 2016-06-08; First posted 2016-09-26 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrophysiological Study (Experimental): Subjects will receive pacing from one right ventricular lead and one left ventricular catheter/lead with multiple LV pacing spots during electrophysiological study procedure.
  Interventions: Procedure: Electrophysiological Study

INTERVENTIONS:
Procedure: Electrophysiological Study — Subjects will receive pacing from one right ventricular lead and one left ventricular catheter/lead with multiple LV pacing spots during electrophysiological study procedure.

SUMMARY:
The SYNSEQ study intends to assess the positive left ventricular dP/dt max achieved by MultiSpot LV pacing (either simultaneously or sequentially) in comparison to the response achieved by the current (standard) BiV pacing configuration in patients indicated/recommended for cardiac resynchronization therapy.

DETAILED DESCRIPTION:
The following pacing configurations will be evaluated.

Biventricular pacing (BiV):

Pacing will be performed on one LV electrode pair, (at 3 different longitudinal locations), and on the tip of the RV-lead. In total, three different pacing BiV settings will be evaluated. Configuration 1: RV + LV lateral Apex, Configuration 2: RV + LV lateral Mid, Configuration 3: RV + LV lateral Base (Reference: Standard CRT)

MultiSpot simultaneous LV-ventricular pacing (MultiSpot-SYN):

Pacing will be performed on 3 electrodes on the LV wall, placed at different longitudinal locations, and on the tip of the RV-lead simultaneously. Configuration 4: RV + LV lateral Apex + LV lateral Mid + LV lateral Base

MultiSpot sequential LV-ventricular pacing (MultiSpot-SEQ):

3 electrodes on the LV wall will be paced sequentially. The RV electrode will be paced simultaneously with last paced LV electrode.The timing-sequence and the amount of spots will depend on the electrical delays measured during the experiments. Configuration 5: LV lateral Apex => LV lateral Mid => LV lateral Base + RV

ELIGIBILITY:
Inclusion Criteria:

* Subject is indicated or recommended for CRT-P or CRT-D device according to current applicable ESC/AHA guidelines
* Subject is in sinus rhythm
* Subject receives optimal heart failure oral medical therapy
* Subject is willing to sign the informed consent form
* Subject is 18 years or older

Exclusion Criteria:

* Subject has permanent atrial fibrillation/flutter or tachycardia
* Subject has pure right bundle branch block (= no additional left ventricular conduction delays)
* Subject has left bundle branch block and QRS-duration of > 150 ms and no sign of myocardial scar indicated by late gadolinium enhancement MRI
* Subject experienced recent myocardial infarction, within 40 days prior to enrollment
* Subject underwent valve surgery, within 90 days prior to enrollment
* Subject is post heart transplantation, or is actively listed on the transplantation list
* Subject is implanted with a left ventricular assist device
* Subject has severe renal disease (up to physicians discretion)
* Subject is on continuous or uninterrupted infusion (inotropic) therapy for heart failure (≥ 2 stable infusions per week)
* Subject has severe aortic stenosis (with a valve area of <1.0 cm2 or significant valve disease expected to be operated within study period)
* Subject has complex and uncorrected congenital heart disease
* Subject has a mechanical heart valve
* Pregnant or breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth control
* Subject is enrolled in another study that could confound the results of this study, without documented pre-approval from Medtronic study manager

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Poland (2):
  - Klinika Choroby Wieńcowej, Warsaw
  - Medical University of Silesia, Silesian Center for Heart Disease,, Zabrze
- Slovakia (2):
  - Národný ústav srdcových a cievnych chorôb, a.s. (NUSCH), Bratislava
  - Východoslovenský ústav srdcových a cievnych chorôb, a.s. (VUSCH), Košice
- Hospital Universitari I Politècnic La Fe, Valencia, Spain
- Skåne University Hospital, Lund, Sweden
- Queen Elizabeth Medical Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sterlinski M, Zakrzewska-Koperska J, Maciag A, Sokal A, Osca-Asensi J, Wang L, Spyropoulou V, Maus B, Lemme F, Okafor O, Stegemann B, Cornelussen R, Leyva F. Acute Hemodynamic Effects of Simultaneous and Sequential Multi-Point Pacing in Heart Failure Patients With an Expected Higher Rate of Sub-response to Cardiac Resynchronization Therapy: Results of Multicenter SYNSEQ Study. Front Cardiovasc Med. 2022 May 12;9:901267. doi: 10.3389/fcvm.2022.901267. eCollection 2022. PMID 35647062

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Electrophysiological Study
Started | 31
Completed | 25 (Subjects who completed electrophysiological study with analyzable data)
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — No veins available for lead placement | 1
Not completed — Electrical instability of patient | 1
Not completed — ECG acquisition error due to sweating | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patient except patient with protocol deviation (subject was not eligible for study)
Arm/Group | Electrophysiological Study
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 1
  Poland | 21
  United Kingdom | 6
  Spain | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Positive Left Ventricular dP/dt Max (mmHG/Sec)
Description: LV dP/dt max is a measurement of the initial velocity of myocardial contraction and is derivative of the LV-pressure. The percentage changes correspond to a percentage change between a pacing configuration (pacing on, e.g., Multispot pacing) and baseline (LV pacing off). There are several repetitions of pacing off and on for each pacing configuration. For one repetition, the percentage change is determined as ([median dP/dt max during pacing On] - (median baseline dP/dt max during pacing Off])/[median dP/dt max during pacing Off]. From all percentage changes for a given pacing configuration and subject, a regression analysis is performed to determine the regression predicted highest percentage change. The presented percentage change is the average over all subjects.
Time Frame: Participants were followed for the time of the EP procedure, which had a median duration of 48 min
Population: The analysis population contains all subjects who completed electrophysiological study with analyzable data. For some patients not all pacing configurations were applied. Two patients missed Multispot sequential pacing and one patient missed BiV mid pacing.
Measure: Mean (Standard Error); unit: % change LV dP/dt max
Arm/Group | Electrophysiological Study
Number analyzed (Participants) | 25
% change LV dP/dt max
  BiV apical | 10.59 (2.56)
  BiV mid: number analyzed (Participants) | 24
  BiV mid | 12.20 (2.06)
  BiV basal | 11.51 (2.15)
  Multispot simultaneous | 15.64 (3.31)
  Multispot sequential: number analyzed (Participants) | 23
  Multispot sequential | 11.80 (2.03)

2. Secondary Outcome: Correlation Between Percentage Change LV dP/dt Max and Percentage Change Blood Pressure
Description: Measured by invasive arterial blood line connected to a sensitive membrane displacement sensor. Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were collected.The percentage changes correspond to a percentage change between a pacing configuration (pacing on, e.g., Multispot pacing) and baseline (LV pacing off). There are several repetitions of pacing off and on for each pacing configuration. For one repetition, the percentage change is determined as ([median pressure during pacing On] - (median pressure during pacing Off])/[median pressure during pacing Off]. Correlation will be summarized over all pacing configurations and time points since the interest is in the overall correlation between LV dP/dt max and other measurements, not in the correlation per pacing configuration or per time point. The general linear model as described in Blank & Altman, Biometrical Journal 310 (1995), p 446, was used to determine the correlation.
Time Frame: Participants were followed for the time of the EP procedure, which had a median duration of 48 min
Population: All patients with analyzable LV dP/dt max data and analyzable and/or available blood pressure data. Two patients of the 25 patients with analyzable LV dP/dt max data did not have blood pressure data available or analyzable.
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Electrophysiological Study
Number analyzed (Participants) | 23
Correlation coefficient
  Correlation between % change LV dP/dt max and SBP | 0.52 [0.50 to 0.54]
  Correlation between % change LV dP/dt max and DBP | 0.37 [0.35 to 0.40]

3. Secondary Outcome: Correlation Between Percentage Change LV dP/dt Max and Percentage Change Non-Invasive Blood Pressure
Description: Acquired through finger volume clamp
Time Frame: Participants were followed for the time of the EP procedure, which had a median duration of 48 min
Population: The collection of non-invasive blood pressures was optional. During study execution, it was decided to not collect and/or analyze any non-invasive blood pressures.
Arm/Group | Electrophysiological Study
Number analyzed (Participants) | 0

4. Secondary Outcome: Correlation Between Percentage Change LV dP/dt Max and Q-LV Ratio
Description: Derived from intra-cardiac leads (invasive) and surface electrodes (non-invasive) respectively. The Q-LV interval is defined as the time from the onset of the QRS width of the surface ECG to the first large positive or negative peak of the LV electrogram (EGM) during a cardiac cycle. The Q-LV ratio will be calculated as Q-LV/QRS duration. Correlation will be summarized over all pacing configurations since the interest is in the overall correlation between LV dP/dt max and other measurements, not in the correlation per pacing configuration. The general linear model as described in Blank & Altman, Biometrical Journal 310 (1995), p 446, was used to determine the correlation between % change LV dP/dt max and Q-LV ratio.
Time Frame: Participants were followed for the time of the EP procedure, which had a median duration of 48 min
Population: The analysis population contains all subjects who completed electrophysiological study with analyzable data. For five patients no Q-LV timings were available for analysis.
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Electrophysiological Study
Number analyzed (Participants) | 20
Correlation coefficient | 0.20 [-0.06 to 0.44]

5. Secondary Outcome: Correlation Between Percentage Change LV dP/dt Max and % Change QRS Width
Description: Derived from surface electrodes (non-invasive). The percentage change is determined as ([QRS width during pacing On] - (QRS width during pacing Off])/[QRS width during pacing Off]. The correlation between % change LV dP/dt max and % change QRS width will be summarized over all pacing configurations since the interest is in the overall correlation between LV dP/dt max and other measurements, not in the correlation per pacing configuration or per time point. The general linear model as described in Blank & Altman, Biometrical Journal 310 (1995), p 446, was used to determine the correlation.
Time Frame: Participants were followed for the time of the EP procedure, which had a median duration of 48 min
Population: The analysis population contains all subjects who completed electrophysiological study with analyzable data. For one patient no QRS width was available for analysis.
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Electrophysiological Study
Number analyzed (Participants) | 24
Correlation coefficient | -0.28 [-0.44 to -0.10]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to study exit. Follow-up time (enrollment to exit) for subjects varied from 1 to 113 days.
Groups:
- Enrolled Subjects: All patients that signed informed consent will be summarized
Arm/Group | Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 3/31
Other Adverse Events (participants affected / at risk) | 2/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=31)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Lead dislogdement (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=31)
Cardiac vein dissection (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-05-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT02914457/SAP_000.pdf
  • Study Protocol (2015-10-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT02914457/Prot_001.pdf